CLINICAL TRIAL: NCT00194194
Title: The Effect of Measuring Resting Metabolic Rate (RMR) in the Context of Moderate or Intensive Behavior Modification Treatment on Weight Loss
Brief Title: Healthetech, Inc. SMART Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: University of Pennsylvania (Other); St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Gary Foster, PhD, Temple University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 801363; NCT00350558 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2008-10

CONDITIONS: Moderate Behavior Management; Intensive Behavior Management
Keywords: BMI; RMR; Personal Computer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- moderate (Active Comparator): moderate behavioral management
  Interventions: Behavioral: moderate
- intensive (Experimental): intensive behavioral management
  Interventions: Device: Resting Metablic Rate measurements

INTERVENTIONS:
Behavioral: moderate — moderate behavioral management with RD
  Other Names: RD
  Arms: moderate
Device: Resting Metablic Rate measurements — intensive behavior management
  Other Names: RMR
  Arms: intensive

SUMMARY:
This study is designed to gain experience with the HealtheTech measurement system (BalanceLog) in the context of a clinical trial and to develop the related treatment protocols. In this study the aim is to evaluate two interventions, one moderate and the other intensive behavioral management. The development and evaluation of a HealtheTech protocol across these two treatment settings will provide useful data about implementation (e.g., technical issues, clinical issues, participant satisfaction) and outcomes (weight loss, retention). These data can provide empirical and clinical support for practice guidelines.

DETAILED DESCRIPTION:
Study Duration: The duration of the study is approximately one year (51 weeks), divided into four phases: 1) Pre-study, 2) Baseline, 3) Intervention, and 4) Maintenance. Participants will be oriented to the procedures and equipment during the pre-study phase (first 3 weeks). During the baseline and intervention phases (24 weeks), participants will be undergoing weight loss treatment. Participants will maintain their weight loss during the maintenance phase (24 weeks).

Subject Recruitment and Selection : Participants will be 80 participants (BMI of 25 to 43 kg/m2) age > 21 years who have access to a personal computer (PC). The anticipated gender balance in the study group will be 80% females and 20% males. Forty participants will be recruited at the University of Pennsylvania and 40 at St. Luke's Hospital in New York City. Participants will be randomly assigned to a moderate or intensive intervention (described below).

Research Design : This study is divided into four phases:

Phase 1 (Pre-study): Screening medical and nutritional evaluation, RMR measurement, Balance Log orientation. There will be 3 weeks in which participants learn how to use the BalanceLog Pro technology, including transferring information to the clinic (i.e., at week -3 become familiar with logging and establish a Balance Log Pro account, log meals and activity and upload data to the Balance Log Pro at week -2, learn how to use special Balance Log functions such as adding foods and receive feedback via email concerning Balance Log Pro upload at week -1). In order to be randomized, participants will need to be proficient in the use of technology so that that treatment can focus on inducing weight loss rather than learning the software.

Phase 2 (Baseline): All participants will participate in weekly individual meetings with the dietitian (R.D.) for 6 weeks. This is designed to establish a solid base for the study and provide a good start on weight loss.

Phase 3 (Intervention): Individuals will be randomized to either a moderate or intensive intervention. Paricipants in the moderate intervention will meet individually with the RD once per month. Individuals in the intensive intervention will meet with the RD twice per month. This Phase continues for 18 weeks - this makes the weight loss phase of the study 6 months in length. A second DEXA scan will be completed at the end of this study phase.

Phase 4 (Maintenance): From 6 to 12 months all participants will shift to a maintenance phase and be contacted and measured at 9 and 12 months. At these timepoints, participants will meet individually with the RD. All individuals use the same HETC tools (MedGem, BalanceLog, and BalanceLog Pro).

Behavioral treatment will be based on the LEARN Program for Weight Control Manual. Participants will be encouraged to consume a low-calorie, low-fat diet (i.e., 30% of calories from fat, 15% of calories from protein and 55% of calories from carbohydrate). The Balance Log, a software tool, will be used to establish a calorie prescription based on a variety of individual factors like RMR, lifestyle activity, and physical activity level as described in the Balance Log software.

1. Moderate Frequency. Participants in this condition will be provided information about the treatment program (LEARN Manual, schedule) and how to use Balance Log (version 2.1.1 and professional web-based program) to log food intake and activity. Participants in this group will meet with a dietitian individually on a weekly basis for the first 6 weeks, then once a month for the remaining 18 weeks of the weight loss phase. During the last 6 months of the study (i.e., weight maintenance phase), participants will meet with a dietitian for quarterly follow-up.
2. Intensive Frequency. Participants in this condition will be provided information about the treatment program (LEARN Manual, schedule) and how to use Balance Log (version 2.1.1 and professional web-based program) to log food intake and activity. Participants in this group will meet with a dietitian individually on a weekly basis for the first 6 weeks, then biweekly for the remaining 18 weeks of the weight loss phase. During the last 6 months of the study (i.e., weight maintenance phase), participants will meet with a dietitian for quarterly follow-up.

Program materials. The materials will be based on the current weight management program at the University of Pennsylvania. Additional materials will be developed or altered to reflect HealtheTech messaging (RMR, energy balance, self-monitoring, etc.). HealtheTech will provide some support for content and layout (graphics and professional reproduction).

A complete set of Program Guideline materials will be developed as a result of the study. The principal investigators will develop materials such as:

• Topical outline of the 20 sessions for clinicians • Talking point summaries for each session • "What to do" summaries for the participants • Skill builders to be used in each session • Key messages sequenced throughout the program

Assessments: The following assessments will be performed:

Blood tests. Routine blood work, including a comprehensive metabolic panel, complete blood count and lipid panel, will be performed during baseline and week 24. Blood samples will be discarded following analysis.

Waist circumference. Waist circumference will be measured at baseline and on weeks 2, 4, 8, 12, 16, 20, 24, 38 and 52. Waist circumference will be measured at the mid-point between the right iliac crest and the bottom of the right rib cage using a Gulick measuring tape.

Body composition. Body composition will be measured by dual x-ray absorptiometry (DEXA) at baseline and week 24. DEXA will provide estimates of total body fat (and fat free mass) and bone mineral density (hip, spine and total body). The body composition unit will be performed at the Children's Hospital of Philadelphia (CHOP) body composition laboratory which is located on 3550 Market, 4th floor. A urine pregnancy test will be given to all women prior to each DEXA scan.

Weight. Weight will be measured at screening, baseline, and at each treatment visit using a digital scale with subjects dressed in light clothing and without shoes. Height will be measured using a stadiometer at screening and at weeks 52 and 104.

Blood Pressure. Blood pressure will be measured at screening, baseline and weeks 2, 4, 8, 12, 16, 20, 24, 38 and 52. On each occasion, two readings will be taken, 1 minute apart after you have been seated for 5 minutes. All measurements will be performed at the WEDP.

Resting Metabolic Rate. The MedGem will be used for all RMR measurements. RMR measurements will be conducted at baseline and weeks 2, 4, 8, 12, 16, 20, 24, 38 and 52. All participants will have their RMR measured once during the pre-study phase to develop familiarization with the test. RMR measurements will be repeated when the opinion of the clinician is there has been a problem or the result is outside of reasonable, Harris-Benedict (the traditional RMR prediction formula) + 15% range. The MINIMUM rate of weight loss will be calculated based on 10% weight loss divided over 24 weeks. (Examples: 240 lb participant: 24 lb weight loss over 24 weeks, 1 lb/week, 500 kcal deficit per day; whereas a 180 lbs. participant would have a target of 18 lbs over the 24 weeks or 0.67 lbs/week or a daily caloric deficit of 367 kcal/day).

Caloric Budget Adjustments Based on RMR: Adjustments to calorie budgets will be done monthly when appropriate. Although we are measuring RMR at week 2, calorie budgets will not be adjusted at this time. The investigators will provide a recommendation for the number of kcal/day that a RMR must change before the Individualized Energy Balance Prescription (IEBP) is recalculated. For example, if there is a 50 kcal/day difference, then it may not be meaningful to change the IEBP, that only represents a change of about 3%, whereas if the change is 150 or more kcal/day it is reasonable to change the recommended intake.

Resting metabolic rate will be measured under strict resting conditions:

12 hour fast (including caffeine) 12 hours post-exercise 30 minute rest prior to the measurement A 2 to 3 minute familiarization will be done with the device during the resting period.

Dietary Intake and Activity. Individuals will be required to log their food and exercise daily for 6 months. They will log using BalanceLog on their PC. One of the inclusion criterions will be daily access to a PC. The BalanceLog will be used to establish an Energy Balance Prescription for all participants. Macronutrient composition will be chosen by the participant, however the recommendation will be to use a relatively standard low (<30 %) fat diet with a minimum of 40% carbohydrate. BalanceLog Pro is a web-based program allowing professionals to review individuals' BalanceLog records and reports remotely.

Questionnaires. A qualitative assessment of logging will be conducted at two time points (3 months and 6 months). Process measures including ease and frequency of use, participant satisfaction, ratings of professional staff.

Potential Risks: The program of weight loss treatment presents few risks to participants. Psychological risks include subjective distress in participants who regain their weight. We will acknowledge participants' disappointment and discuss their experiences from the perspectives of others who have regained weight.

The potential risks of the study are primarily associated with the assessment measures, specifically the DEXA and blood testing. The blood tests present a minor risk of bruising. Every effort will be made to minimize these risks including a review of participants' health before the testing.

Informed Consent : Participants will be recruited from public service announcements, notices in local newspapers, and referrals from physicians' offices at the three sites. Applicants will be screened by phone to determine that they meet the recruitment criteria, have no obvious contraindications to treatment, and remain interested in the study after it has been described. Screenings will be conducted by research coordinators following a written protocol. Persons who appear appropriate to participate will be scheduled for an initial interview. In the face-to-face interview, applicants will be informed of the nature and requirements of the study, including randomization to treatment conditions. They will be provided a written description of all study details and asked to give their informed consent to participate in further assessment and treatment. Candidates not wishing to participate, or who do not meet criteria, will be offered a referral to an appropriate program.

Protection of Participants: Risks of complications will be reduced by carefully selecting participants for treatment. We have clearly defined the contraindications and will inform the participants' primary care physicians of these contraindications. Participants will receive blood tests at frequent intervals, and results of these tests will be monitored by a physician to ensure participant safety during weight loss. Both participants and their primary care physicians will be made aware of any abnormal findings.

Data will be kept in a locked file cabinet to ensure confidentiality. In addition, guidelines concerning the confidentiality of group treatment sessions will be reviewed with participants at the initial interview and at the first treatment session. Code numbers will be assigned to each participant to maximize anonymity while entering data.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 to 43 kg/m2
* age > 21 years
* access to a personal computer (PC)

Exclusion Criteria:

* BMI above/below 25-43 kg/m2
* age < 21 years
* no access to a personal computer (PC)
* type 2 diabetes
* participants taking medications known to affect weight, appetite or energy expenditure

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2004-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
This study is designed to gain experience with the HealtheTech measurement system (BalanceLog) in the context of a clinical trial and to develop the related treatment protocols | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foster, Ph.D., Principal Investigator — Temple University - Center for Obesity Research and Education; Steven B Heymsfield, M.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Temple University- Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States